CLINICAL TRIAL: NCT03002402
Title: Feasibility and Acceptability of an Internet-based Cognitive-behavioral Treatment for Insomnia in Adults With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Faith Luyster, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R03HL135213-01 (NIH); 1R03HL135213-01 (NIH)
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Asthma; Insomnia Chronic
Keywords: asthma; insomnia; cognitive-behavioral treatment
MeSH Terms: conditions — Asthma; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-based CBT-I (Experimental): Sleep Healthy Using the Internet (SHUTi) is a self-guided, automated, interactive, and tailored web-based program modeled on the primary tenets of cognitive-behavioral treatment for insomnia (CBT-I): sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention. Intervention content is allocated out over time through 6 "Cores." Users obtain access to a new Core based on a time and event-based schedule (e.g., 7 days after completion of previous Core). SHUTi uses online sleep diaries to track progress and to tailor treatment (e.g., assign a sleep restriction window).
  Interventions: Behavioral: Internet-based CBT-I

INTERVENTIONS:
Behavioral: Internet-based CBT-I — Internet-based cognitive-behavioral treatment for insomnia
  Other Names: Sleep Healthy Using the Internet (SHUTi)

SUMMARY:
The purpose of the proposed study are to explore changes in sleep and asthma outcomes from baseline to post-treatment in adults with asthma and comorbid insomnia who underwent Internet-based cognitive-behavioral treatment for insomnia (CBT-I).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of moderate-severe persistent asthma
* Not well controlled asthma (score ≤ 19 on the Asthma Control Test)
* Age 18-75 years
* Meets criteria for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Insomnia Disorder
* At least moderate insomnia severity (score ≥ 10 on Insomnia Severity Index)
* Telephone number, email address, and reliable Internet access

Exclusion Criteria:

* History of bipolar or psychosis
* Substance abuse disorder within past 3 months
* Dementia or probable dementia diagnosis
* Plans to move or leave present source of care during the following 6 months.
* Non-English speaking, illiterate, or possesses sensory deficits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | baseline and post-intervention (up to 9 weeks)
  Insomnia Severity Index
Asthma control | baseline and post-intervention (up to 9 weeks)
  Asthma Control Test

CONTACTS AND LOCATIONS:
Overall Officials: Faith S Luyster, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No